CLINICAL TRIAL: NCT00493285
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation Study to Evaluate the Safety, Tolerability,Immunogenicity, and Viral Shedding of MEDI-534, a Live, Attenuated Intranasal Vaccine Against Respiratory Syncytial Virus (RSV) and Parainfluenza Virus Type 3 (PIV), in Healthy Children 6 to <24 Months of Age
Brief Title: Safety and Tolerability Study to Evaluate MEDI-534 in Children 6 to < 24 Months of Age
Acronym: CP149
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Elissa Malkin, D.O., MedImmune LLC
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MI-CP149
Record Dates: First submitted 2007-06-26; First posted 2007-06-28 (Estimated); Results first posted 2012-04-09 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: Respiratory Viral Infections; Respiratory Syncytial Virus Infections; Parainfluenza Virus 3, Human
Keywords: Lower Respiratory Tract Illness; RSV and PIV3 infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): MEDI-534 at 10^4 TCID50 at 0, 2, and 4 months (Nasal spray)
  Interventions: Biological: MEDI-534
- 2 (Active Comparator): MEDI-534 at 10^5 TCID50 at 0, 2, and 4 months (Nasal Spray)
  Interventions: Biological: MEDI-534
- 3 (Active Comparator): MEDI-534 at 10^6 TCID50 at 0, 2, and 4 months (Nasal Spray)
  Interventions: Biological: MEDI-534

INTERVENTIONS:
Biological: MEDI-534 — Multiple doses of MEDI-534 or Placebo at 10^4 TCID50
  Arms: 1
Biological: MEDI-534 — Multiple doses of MEDI-534 or Placebo at 10 ^5 TCID50.
  Arms: 2
Biological: MEDI-534 — Multiple doses of MEDI-534 or Placebo at 10^6 TCID50.
  Arms: 3

SUMMARY:
The overall objective of the MEDI-534 clinical development program is to evaluate the safety, efficacy and tolerability of MEDI-534 for the prevention of serious RSV and PIV3 disease in young infants.

DETAILED DESCRIPTION:
The primary objective of this study is to describe the safety and tolerability of multiple doses of MEDI-534 at 10^4, 10^5, or 10^6 TCID50 when administered to RSV and PIV3 seronegative children 6 to <24 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Male or female whose age on the day of randomization is 6 to <24 months (reached 6th month birthday and not yet reached 2nd year birthday)
* Subject is seronegative to both RSV and PIV3 at screening
* Subject was the product of normal full term pregnancy (defined as >36 weeks gestation)
* Subject is in general good health
* Subject's legal representative is available by telephone
* Written informed consent and HIPAA authorization (if applicable) obtained from the subject's legal representative
* Subject's legal representative is able to understand and comply with the requirements of the protocol as judged by the investigator
* Subject is available to complete the follow-up period, which will be through the end of RSV season (provisionally defined as 01/Apr for the United States) or 180 days after the final dose of study vaccine, whichever is later
* Subject's legal representative must be willing and able to bring the subject to the study site for evaluation of respiratory illness in accordance with the protocol

Exclusion Criteria:

* Any fever (equal to or greater than 100.4°F [equal to or greater than 38.0°C], regardless of route) or lower respiratory illness (Section 4.1.2) within 7 days prior to randomization
* Moderate or severe nasal congestion that in the investigator's opinion could prevent intranasal delivery of vaccine
* Any drug therapy (chronic or other) within 7 days prior to randomization or expected receipt through the protocol-specified blood collection 28 days after each study vaccine dosing, except that infrequent use of over-the-counter medications such as pain relievers are permitted according to the judgment of the investigator
* Any current or expected receipt of immunosuppressive agents including steroids (2 mg/kg per day of prednisone or its equivalent, or equal to or greater than 20 mg/day if the subject weighs >10 kg, given daily or on alternate days for equal to or greater than 14 days); children in this category should not receive study vaccine until immunosuppressive agents including corticosteroid therapy have been discontinued for equal to or greater than 30 days; the use of topical steroids is permitted according to the judgment of the investigator
* History of receipt of blood transfusion or expected receipt through 30 days following final study vaccine dosing
* History of receipt of immunoglobulin products or expected receipt through 30 days after study vaccine dosing
* Receipt of any investigational drug within 60 days prior to randomization or expected receipt through 30 days after final study vaccine dosing
* Receipt of any live virus vaccine (excluding rotavirus vaccine) within 28 days prior to randomization or expected receipt within a 28-day window around any study vaccine dose
* Receipt of any inactivated (i.e., non-live) vaccine or rotavirus vaccine within 14 days prior to randomization or expected receipt within a 14-day window around any study vaccine dose
* Known or suspected immunodeficiency, including HIV
* Living in the same home or enrolled in the same classroom at day care with infants <24 months of age (only one child per household may be enrolled into the study)
* Contact with pregnant caregiver
* A household contact who is immunocompromised; the subject should also avoid close contact with immunocompromised individuals for at least 30 days after any study vaccine dose
* A household contact who is a health care provider in contact with immunocompromised patients or who is a day care provider for infants under the age of 6 months
* History of allergic reaction to any component of the study vaccine
* Previous medical history, or evidence, of an intercurrent or chronic illness that, in the opinion of the investigator, may compromise the safety of the subject
* Known or suspected active or chronic hepatitis infection
* History of medical diagnosis of asthma, reactive airway disease, wheezing requiring medication, cystic fibrosis, bronchopulmonary dysplasia, chronic pulmonary disease, medically confirmed apnea, hospitalization for respiratory illness or mechanical ventilation
* Family member or household contact who is an employee of the research center or otherwise involved with the conduct of the study
* Any condition that, in the opinion of the investigator, might interfere with study vaccine evaluation

Ages: 6 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2007-07; Primary Completion 2009-11 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elissa Malkin, D.O., Study Director — MedImmune LLC
Locations (30):
- United States (30):
  - Arkansas Pediatric Research Division, Conway, Arkansas
  - Arkansas Pediatric Clinic, Little Rock, Arkansas
  - THe Children's Hospital, Aurora, Colorado
  - Miami Children's Hospital, Miami, Florida
  - Pediatric Partners, Palm Beach Gardens, Florida
  - North Georgia Clinical Research Center, Dalton, Georgia
  - University Consultants in Allergy and Immunology, Chicago, Illinois
  - Children's Memorial Hospital, Chicago, Illinois
  - University of Maryland, Baltimore, Baltimore, Maryland
  - Tufts-New England Medical Center, Boston, Massachusetts
  - Craig A. Spiegel, MD, Bridgeton, Missouri
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - United Medical Associates, Binghamton, New York
  - Withrop University Hospital, Mineola, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University Hospitals case Medical Center, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - St. Vincent Mercy Medical Center Mercy Children's Hospital, Toledo, Ohio
  - Primary Physicians Research, Inc., Pittsburgh, Pennsylvania
  - Sanford Children's Specialty Clinic, Sioux Falls, South Dakota
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Health Science Center of Houston Medical School, Houston, Texas
  - Bear Care Pediatrics, Ogden, Utah
  - Copperview Medical Center, South Jordan, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - Advanced Pediatrics, Vienna, Virginia
  - Rockwood Clinic Research Center, Spokane, Washington
  - Marshall University Joan C. Edwards School of Medicine, Huntington, West Virginia
  - West Virginia University Health Science Center, Morgantown, West Virginia

REFERENCES:
- [Result] Bernstein DI, Malkin E, Abughali N, Falloon J, Yi T, Dubovsky F; MI-CP149 Investigators. Phase 1 study of the safety and immunogenicity of a live, attenuated respiratory syncytial virus and parainfluenza virus type 3 vaccine in seronegative children. Pediatr Infect Dis J. 2012 Feb;31(2):109-14. doi: 10.1097/INF.0b013e31823386f1. PMID 21926667

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants 6 to < 24 months of age were screened prior to randomization at 13 sites in the USA. The first subject entered the study on 02Jul2007 and the last subject completed the study on 20Apr2010.
Pre-assignment Details: A total of 49 participants were entered into the study between 02Jul2007 and 25Jun2009. Participants were RSV and PIV3 seronegative at screening, and randomized in a 2:1 ratio to receive MEDI-534 or placebo, and randomization was stratified by age (≤ 12 months vs > 12 months).
Period: Overall Study
Arm/Group | 10^4 MEDI-534 | 10^4 PLACEBO | 10^5 MEDI-534 | 10^5 PLACEBO | 10^6 MEDI-534 | 10^6 PLACEBO
Started | 13 | 6 | 9 | 6 | 10 | 5
Completed | 13 | 6 | 9 | 6 | 9 | 5
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- TOTAL: Total of all reporting groups
Arm/Group | 10^4 MEDI-534 | 10^4 PLACEBO | 10^5 MEDI-534 | 10^5 PLACEBO | 10^6 MEDI-534 | 10^6 PLACEBO | TOTAL
Number analyzed (Participants) | 13 | 6 | 9 | 6 | 10 | 5 | 49
Age Continuous [Mean (Standard Deviation); unit: Months] | 10.8 (5.0) | 12.2 (7.6) | 8.1 (1.8) | 11.3 (3.7) | 9.3 (2.1) | 9.9 (4.3) | 10.1 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 2 | 5 | 4 | 6 | 3 | 28
  Male | 5 | 4 | 4 | 2 | 4 | 2 | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Adverse Events (SEs) After Dose 1
Description: The SEs for this study included fever ≥ 100.4°F, runny/stuffy nose, cough, drowsiness, loss of appetite/decreased urine output, irritability/fussiness, laryngitis, and epistaxis.
Time Frame: Days 0-28 after Dose 1 (Dose 1 was on Day 0)
Population: Safety population for solicited symptoms included randomized participants who received investigational product for the specified dose and had any solicited symptom data obtained after that dose
Measure: Number; unit: participants
Groups:
- 10^4 MEDI-534; 10^5 MEDI-534; 10^6 MEDI-534: MEDI-534 vaccine was supplied as a frozen preparation of live, attenuated, b/h PIV3/RSV F2 virus filled into syringes. Each 0.2 mL dose contained MEDI-534 in a sucrose phosphate buffer.
- 10^4 Placebo; 10^5 Placebo; 10^6 Placebo: Placebo was supplied as a frozen preparation filled into syringes. Each 0.2 mL dose contained sucrose phosphate buffer.
Arm/Group | 10^4 MEDI-534 | 10^4 Placebo | 10^5 MEDI-534 | 10^5 Placebo | 10^6 MEDI-534 | 10^6 Placebo
Number analyzed (Participants) | 13 | 6 | 9 | 6 | 10 | 5
participants | 12 | 5 | 8 | 6 | 9 | 4

2. Primary Outcome: Number of Participants With SEs After Dose 2
Description: as for outcome 1
Time Frame: Days 0-28 after Dose 2 (Dose 2 was on Day 48-64)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | 10^4 MEDI-534 | 10^4 Placebo | 10^5 MEDI-534 | 10^5 Placebo | 10^6 MEDI-534 | 10^6 Placebo
Number analyzed (Participants) | 11 | 5 | 7 | 6 | 9 | 5
participants | 9 | 5 | 6 | 6 | 6 | 3

3. Primary Outcome: Number of Participants With SEs After Dose 3
Description: as for outcome 1
Time Frame: Days 0-28 after Dose 3 (Dose 3 was 48-64 days after Dose 2)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | 10^4 MEDI-534 | 10^4 Placebo | 10^5 MEDI-534 | 10^5 Placebo | 10^6 MEDI-534 | 10^6 Placebo
Number analyzed (Participants) | 11 | 5 | 5 | 6 | 9 | 5
participants | 9 | 5 | 4 | 5 | 8 | 2

4. Primary Outcome: Number of Participants With Adverse Events (AEs) After Dose 1
Description: Unsolicited AEs reported by 1 or more participants in either treatment group through 28 days post Dose 1.
Time Frame: Days 0-28 after Dose 1 (Dose 1 was on Day 0)
Population: The safety population for AEs included randomized participants who received investigational product for the specified dose and had any safety follow-up.
Measure: Number; unit: participants
Arm/Group | 10^4 MEDI-534 | 10^4 Placebo | 10^5 MEDI-534 | 10^5 Placebo | 10^6 MEDI-534 | 10^6 Placebo
Number analyzed (Participants) | 13 | 6 | 9 | 6 | 10 | 5
participants | 8 | 4 | 8 | 5 | 5 | 3

5. Primary Outcome: Number of Participants With AEs After Dose 2
Description: Unsolicited AEs reported by 1 or more participants in either treatment group through 28 days post Dose 2.
Time Frame: Days 0-28 after Dose 2 (Dose 2 was on Day 48-64)
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | 10^4 MEDI-534 | 10^4 Placebo | 10^5 MEDI-534 | 10^5 Placebo | 10^6 MEDI-534 | 10^6 Placebo
Number analyzed (Participants) | 11 | 5 | 7 | 6 | 9 | 5
participants | 6 | 4 | 5 | 4 | 3 | 2

6. Primary Outcome: Number of Participants With AEs After Dose 3
Description: Unsolicited AEs reported by 1 or more participants in either treatment group through 28 days post Dose 3.
Time Frame: Days 0-28 after Dose 3 (Dose 3 was 48-64 days after Dose 2)
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | 10^4 MEDI-534 | 10^4 Placebo | 10^5 MEDI-534 | 10^5 Placebo | 10^6 MEDI-534 | 10^6 Placebo
Number analyzed (Participants) | 11 | 5 | 5 | 6 | 9 | 5
participants | 7 | 3 | 3 | 3 | 4 | 2

7. Primary Outcome: Number of Subjects With Medically-attended Lower Respiratory Illnesses (MA-LRIs)
Description: An MA-LRI was a healthcare provider-confirmed diagnosis of 1 or more of the following: wheezing, pneumonia, croup, rhonchi (not cleared with cough or suctioning), rales, bronchitis, bronchiolitis, apnea.
Time Frame: Days 0 to 180 days after final dose or the end of the RSV season, whichever was later
Population: The safety population for MA-LRIs included randomized participants who received investigational product and had any safety follow-up.
Measure: Number; unit: participants
Arm/Group | 10^4 MEDI-534 | 10^4 Placebo | 10^5 MEDI-534 | 10^5 Placebo | 10^6 MEDI-534 | 10^6 Placebo
Number analyzed (Participants) | 13 | 6 | 9 | 6 | 10 | 5
participants | 3 | 2 | 2 | 3 | 2 | 1

8. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: Events resulting in death; were life-threatening; resulted in inpatient hospitalization/prolongation of hospitalization; resulted in persistent or significant disability or incapacity; were a congenital anomaly/birth defect in the offspring of a participant; or were an important medical event that may not have resulted in death, threatened life, or required hospitalization and may have jeopardized the participant and required medical/surgical intervention to prevent one of the above outcomes.
Time Frame: Days 0-28 after any dose
Population: The safety population included all subjects who received investigational product for the specified dose and had any safety follow-up.
Measure: Number; unit: participants
Arm/Group | 10^4 MEDI-534 | 10^4 Placebo | 10^5 MEDI-534 | 10^5 Placebo | 10^6 MEDI-534 | 10^6 Placebo
Number analyzed (Participants) | 13 | 6 | 9 | 6 | 10 | 5
participants | 0 | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Participants With Significant New Medical Conditions (SNMCs)
Description: A SNMC is a newly diagnosed medical condition that is of a chronic, ongoing nature and is assessed by the investigator as medically significant.
Time Frame: Day 0 through 180 days after the final dose or through the end of the RSV season, whichever was later
Population: Safety population was participants who received investigational product and had any safety follow-up for ≥ 1 day after dosing (ie, did not discontinue on Day 0 after receiving Dose 1).
Measure: Number; unit: participants
Arm/Group | 10^4 MEDI-534 | 10^4 Placebo | 10^5 MEDI-534 | 10^5 Placebo | 10^6 MEDI-534 | 10^6 Placebo
Number analyzed (Participants) | 13 | 6 | 9 | 6 | 10 | 5
participants | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants Shedding Vaccine-like Virus at Any Time During Study Participation
Description: Number of participants with nasal wash specimens that were positive for RSV or PIV3 by culture and identified as vaccine-type virus by RT-PCR.
Time Frame: Days 7, 12, and 28 after each dose and during visits for pre-specified illness symptoms occurring Day 0 through 28-34 days post each dose.
Population: The shedding population included all subjects who received investigational product and had any valid shedding data.
Measure: Number; unit: participants
Arm/Group | 10^4 MEDI-534 | 10^4 Placebo | 10^5 MEDI-534 | 10^5 Placebo | 10^6 MEDI-534 | 10^6 Placebo
Number analyzed (Participants) | 13 | 6 | 8 | 6 | 10 | 5
participants | 6 | NA — Nasal wash samples from participants receiving placebo were not analyzed for vaccine-type virus shedding. | 5 | NA — Nasal wash samples from participants receiving placebo were not analyzed for vaccine-type virus shedding. | 7 | NA — Nasal wash samples from participants receiving placebo were not analyzed for vaccine-type virus shedding.

11. Secondary Outcome: Number of Participants Shedding Vaccine-like Virus at 7 Days After Dose 1
Description: as for outcome 10
Time Frame: Days 7-10 after Dose 1 (Dose 1 was on Day 0)
Population: The shedding population included all subjects who received investigational product and had any valid shedding data.
Measure: Number; unit: participants
Arm/Group | 10^4 MEDI-534 | 10^4 Placebo | 10^5 MEDI-534 | 10^5 Placebo | 10^6 MEDI-534 | 10^6 Placebo
Number analyzed (Participants) | 13 | 6 | 7 | 6 | 9 | 5
participants | 6 | NA — Nasal wash samples from participants receiving placebo were not analyzed for vaccine-type virus shedding. | 5 | NA — Nasal wash samples from participants receiving placebo were not analyzed for vaccine-type virus shedding. | 6 | NA — Nasal wash samples from participants receiving placebo were not analyzed for vaccine-type virus shedding.

12. Secondary Outcome: Number of Participants Shedding Vaccine-like Virus at 12 Days After Dose 1
Description: as for outcome 10
Time Frame: Days 12-18 after Dose 1 (Dose 1 was on Day 0)
Population: The shedding population included all subjects who received investigational product and had any valid shedding data.
Measure: Number; unit: participants
Arm/Group | 10^4 MEDI-534 | 10^4 Placebo | 10^5 MEDI-534 | 10^5 Placebo | 10^6 MEDI-534 | 10^6 Placebo
Number analyzed (Participants) | 13 | 6 | 8 | 6 | 10 | 5
participants | 1 | NA — Nasal wash samples from participants receiving placebo were not analyzed for vaccine-type virus shedding. | 3 | NA — Nasal wash samples from participants receiving placebo were not analyzed for vaccine-type virus shedding. | 2 | NA — Nasal wash samples from participants receiving placebo were not analyzed for vaccine-type virus shedding.

13. Secondary Outcome: Number of Participants Shedding Vaccine-like Virus at 28 Days After Dose 1
Description: as for outcome 10
Time Frame: Days 28-34 after Dose 1 (Dose 1 was on Day 0)
Population: The shedding population included all subjects who received investigational product and had any valid shedding data.
Measure: Number; unit: participants
Arm/Group | 10^4 MEDI-534 | 10^4 Placebo | 10^5 MEDI-534 | 10^5 Placebo | 10^6 MEDI-534 | 10^6 Placebo
Number analyzed (Participants) | 13 | 6 | 7 | 6 | 9 | 5
participants | 0 | NA — Nasal wash samples from participants receiving placebo were not analyzed for vaccine-type virus shedding. | 0 | NA — Nasal wash samples from participants receiving placebo were not analyzed for vaccine-type virus shedding. | 0 | NA — Nasal wash samples from participants receiving placebo were not analyzed for vaccine-type virus shedding.

14. Secondary Outcome: Number of Participants With Shedding of Vaccine-like Virus on Any Day During Days 0-28 After Dose 1
Description: as for outcome 10
Time Frame: Days 0-34 after Dose 1 (Dose 1 was on Day 0)
Population: The shedding population included all subjects who received investigational product and had any valid shedding data.
Measure: Number; unit: participants
Arm/Group | 10^4 MEDI-534 | 10^4 Placebo | 10^5 MEDI-534 | 10^5 Placebo | 10^6 MEDI-534 | 10^6 Placebo
Number analyzed (Participants) | 13 | 6 | 8 | 6 | 10 | 5
participants | 6 | NA — Nasal wash samples from participants receiving placebo were not analyzed for vaccine-type virus shedding. | 5 | NA — Nasal wash samples from participants receiving placebo were not analyzed for vaccine-type virus shedding. | 7 | NA — Nasal wash samples from participants receiving placebo were not analyzed for vaccine-type virus shedding.

15. Secondary Outcome: Number of Participants Shedding Vaccine-like Virus at 7 Days After Dose 2
Description: as for outcome 10
Time Frame: Days 7-10 after Dose 2 (Dose 2 was on Day 48-64)
Population: The shedding population included all subjects who received investigational product and had any valid shedding data.
Measure: Number; unit: participants
Arm/Group | 10^4 MEDI-534 | 10^4 Placebo | 10^5 MEDI-534 | 10^5 Placebo | 10^6 MEDI-534 | 10^6 Placebo
Number analyzed (Participants) | 9 | 6 | 7 | 6 | 8 | 5
participants | 0 | NA — Nasal wash samples from participants receiving placebo were not analyzed for vaccine-type virus shedding. | 1 | NA — Nasal wash samples from participants receiving placebo were not analyzed for vaccine-type virus shedding. | 0 | NA — Nasal wash samples from participants receiving placebo were not analyzed for vaccine-type virus shedding.

16. Secondary Outcome: Number of Participants Shedding Vaccine-like Virus at 12 Days After Dose 2
Description: as for outcome 10
Time Frame: Days 12-18 after Dose 2 (Dose 2 was on Day 48-64)
Population: The shedding population included all subjects who received investigational product and had any valid shedding data.
Measure: Number; unit: participants
Arm/Group | 10^4 MEDI-534 | 10^4 Placebo | 10^5 MEDI-534 | 10^5 Placebo | 10^6 MEDI-534 | 10^6 Placebo
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 9 | 5
participants | 0 | NA — Nasal wash samples from participants receiving placebo were not analyzed for vaccine-type virus shedding. | 0 | NA — Nasal wash samples from participants receiving placebo were not analyzed for vaccine-type virus shedding. | 0 | NA — Nasal wash samples from participants receiving placebo were not analyzed for vaccine-type virus shedding.

17. Secondary Outcome: Number of Participants Shedding Vaccine-like Virus at 28 Days After Dose 2
Description: as for outcome 10
Time Frame: Days 28-34 after Dose 2 (Dose 2 was on Day 48-64)
Population: The shedding population included all subjects who received investigational product and had any valid shedding data.
Measure: Number; unit: participants
Arm/Group | 10^4 MEDI-534 | 10^4 Placebo | 10^5 MEDI-534 | 10^5 Placebo | 10^6 MEDI-534 | 10^6 Placebo
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 9 | 5
participants | 0 | NA — Nasal wash samples from participants receiving placebo were not analyzed for vaccine-type virus shedding. | 0 | NA — Nasal wash samples from participants receiving placebo were not analyzed for vaccine-type virus shedding. | 0 | NA — Nasal wash samples from participants receiving placebo were not analyzed for vaccine-type virus shedding.

18. Secondary Outcome: Number of Participants With Shedding of Vaccine-like Virus on Any Day During Days 0-28 After Dose 2
Description: as for outcome 10
Time Frame: Days 0-34 after Dose 2 (Dose 2 was on Day 48-64)
Population: The shedding population included all subjects who received investigational product and had any valid shedding data.
Measure: Number; unit: participants
Arm/Group | 10^4 MEDI-534 | 10^4 Placebo | 10^5 MEDI-534 | 10^5 Placebo | 10^6 MEDI-534 | 10^6 Placebo
Number analyzed (Participants) | 11 | 6 | 7 | 6 | 9 | 5
participants | 0 | NA — Nasal wash samples from participants receiving placebo were not analyzed for vaccine-type virus shedding. | 1 | NA — Nasal wash samples from participants receiving placebo were not analyzed for vaccine-type virus shedding. | 0 | NA — Nasal wash samples from participants receiving placebo were not analyzed for vaccine-type virus shedding.

19. Secondary Outcome: Number of Participants Shedding Vaccine-like Virus at 7 Days After Dose 3
Description: as for outcome 10
Time Frame: Days 7-10 after Dose 3 (Dose 3 was 48-64 days after Dose 2)
Population: The shedding population included all subjects who received investigational product and had any valid shedding data.
Measure: Number; unit: participants
Arm/Group | 10^4 MEDI-534 | 10^4 Placebo | 10^5 MEDI-534 | 10^5 Placebo | 10^6 MEDI-534 | 10^6 Placebo
Number analyzed (Participants) | 10 | 6 | 5 | 6 | 9 | 5
participants | 0 | NA — Nasal wash samples from participants receiving placebo were not analyzed for vaccine-type virus shedding. | 0 | NA — Nasal wash samples from participants receiving placebo were not analyzed for vaccine-type virus shedding. | 1 | NA — Nasal wash samples from participants receiving placebo were not analyzed for vaccine-type virus shedding.

20. Secondary Outcome: Number of Participants Shedding Vaccine-like Virus at 12 Days After Dose 3
Description: as for outcome 10
Time Frame: Days 12-18 after Dose 3 (Dose 3 was 48-64 days after Dose 2)
Population: The shedding population included all subjects who received investigational product and had any valid shedding data.
Measure: Number; unit: participants
Arm/Group | 10^4 MEDI-534 | 10^4 Placebo | 10^5 MEDI-534 | 10^5 Placebo | 10^6 MEDI-534 | 10^6 Placebo
Number analyzed (Participants) | 11 | 6 | 5 | 6 | 9 | 5
participants | 0 | NA — Nasal wash samples from participants receiving placebo were not analyzed for vaccine-type virus shedding. | 0 | NA — Nasal wash samples from participants receiving placebo were not analyzed for vaccine-type virus shedding. | 1 | NA — Nasal wash samples from participants receiving placebo were not analyzed for vaccine-type virus shedding.

21. Secondary Outcome: Number of Participants Shedding Vaccine-like Virus at 28 Days After Dose 3
Description: as for outcome 10
Time Frame: Days 28-34 after Dose 3 (Dose 3 was 48-64 days after Dose 2)
Population: The shedding population included all subjects who received investigational product and had any valid shedding data.
Measure: Number; unit: participants
Arm/Group | 10^4 MEDI-534 | 10^4 Placebo | 10^5 MEDI-534 | 10^5 Placebo | 10^6 MEDI-534 | 10^6 Placebo
Number analyzed (Participants) | 10 | 6 | 5 | 6 | 8 | 5
participants | 0 | NA — Nasal wash samples from participants receiving placebo were not analyzed for vaccine-type virus shedding. | 0 | NA — Nasal wash samples from participants receiving placebo were not analyzed for vaccine-type virus shedding. | 0 | NA — Nasal wash samples from participants receiving placebo were not analyzed for vaccine-type virus shedding.

22. Secondary Outcome: Number of Participants With Shedding of Vaccine-like Virus on Any Day During Days 0-28 After Dose 3
Description: as for outcome 10
Time Frame: Days 0-34 after Dose 3 (Dose 3 was 48-64 days after Dose 2)
Population: The shedding population included all subjects who received investigational product and had any valid shedding data.
Measure: Number; unit: participants
Arm/Group | 10^4 MEDI-534 | 10^4 Placebo | 10^5 MEDI-534 | 10^5 Placebo | 10^6 MEDI-534 | 10^6 Placebo
Number analyzed (Participants) | 11 | 6 | 5 | 6 | 9 | 5
participants | 0 | NA — Nasal wash samples from participants receiving placebo were not analyzed for vaccine-type virus shedding. | 0 | NA — Nasal wash samples from participants receiving placebo were not analyzed for vaccine-type virus shedding. | 1 | NA — Nasal wash samples from participants receiving placebo were not analyzed for vaccine-type virus shedding.

23. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum Antibodies to RSV at Baseline
Description: Pre-dose GMT of serum antibody response to RSV as measured by microneutralization assay. Limit of quantification is 5. For results reported as < 5, a value of 2.5 was imputed.
Time Frame: Baseline (Day 0 prior to Dose 1)
Population: The immunogenicity population included all subjects who received investigational product and had valid results from serum samples obtained for immunogenicity evaluation for PIV3 and/or RSV.
Measure: Mean (95% Confidence Interval); unit: GMT
Arm/Group | 10^4 MEDI-534 | 10^4 Placebo | 10^5 MEDI-534 | 10^5 Placebo | 10^6 MEDI-534 | 10^6 Placebo
Number analyzed (Participants) | 13 | 6 | 8 | 5 | 10 | 5
GMT | 14.52 [8.1 to 26.1] | 17.82 [7.9 to 44.9] | 15.42 [10.0 to 23.8] | 3.79 [2.9 to 5.0] | 6.60 [3.8 to 11.5] | 7.58 [3.8 to 17.4]

24. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum Antibodies to RSV at Day 28 Post Dose 1
Description: Post dose GMT of serum antibody response to RSV as measured by microneutralization assay. Limit of quantification is 5. For results reported as < 5, a value of 2.5 was imputed.
Time Frame: Day 28-34 after Dose 1 (Dose 1 was on Day 0)
Population: as for outcome 23
Measure: Mean (95% Confidence Interval); unit: GMT
Arm/Group | 10^4 MEDI-534 | 10^4 Placebo | 10^5 MEDI-534 | 10^5 Placebo | 10^6 MEDI-534 | 10^6 Placebo
Number analyzed (Participants) | 11 | 5 | 7 | 5 | 9 | 5
GMT | 12.08 [6.4 to 24.2] | 10.00 [5.0 to 17.4] | 80.00 [22.1 to 320.0] | 8.71 [2.9 to 40.0] | 29.39 [7.3 to 127.0] | 7.58 [3.8 to 13.2]

25. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum Antibodies to RSV at Day 28 Post Dose 2
Description: as for outcome 24
Time Frame: Day 28-34 after Dose 2 (Dose 2 was on Day 48-64)
Population: as for outcome 23
Measure: Mean (95% Confidence Interval); unit: GMT
Arm/Group | 10^4 MEDI-534 | 10^4 Placebo | 10^5 MEDI-534 | 10^5 Placebo | 10^6 MEDI-534 | 10^6 Placebo
Number analyzed (Participants) | 10 | 5 | 5 | 6 | 9 | 5
GMT | 13.20 [5.4 to 37.6] | 3.79 [2.9 to 5.0] | 22.97 [10.0 to 69.6] | 7.07 [2.8 to 25.2] | 18.52 [8.6 to 43.2] | 5.00 [3.3 to 7.6]

26. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum Antibodies to RSV at Day 28 Post Dose 3
Description: as for outcome 24
Time Frame: Day 28-34 after Dose 3 (Dose 3 was 48-64 days after Dose 2)
Population: as for outcome 23
Measure: Mean (95% Confidence Interval); unit: GMT
Arm/Group | 10^4 MEDI-534 | 10^4 Placebo | 10^5 MEDI-534 | 10^5 Placebo | 10^6 MEDI-534 | 10^6 Placebo
Number analyzed (Participants) | 8 | 4 | 5 | 5 | 8 | 4
GMT | 30.84 [5.5 to 174.5] | 10.00 [2.5 to 160.0] | 22.97 [6.6 to 91.9] | 6.60 [2.9 to 23.0] | 15.42 [7.1 to 33.6] | 3.54 [2.5 to 5.0]

27. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum Hemagglutination Inhibition (HAI) Antibodies to PIV3 at Baseline
Description: Post dose GMT of serum antibody response to PIV3 as measured by HAI assay. Limit of quantification is 4. For results reported as < 4, a value of 2 was imputed.
Time Frame: Baseline (Day 0 prior to Dose 1)
Population: as for outcome 23
Measure: Mean (95% Confidence Interval); unit: GMT
Arm/Group | 10^4 MEDI-534 | 10^4 Placebo | 10^5 MEDI-534 | 10^5 Placebo | 10^6 MEDI-534 | 10^6 Placebo
Number analyzed (Participants) | 13 | 6 | 8 | 5 | 10 | 5
GMT | 3.23 [2.2 to 5.0] | 2.52 [2.0 to 4.0] | 2.59 [2.0 to 4.4] | 4.59 [2.0 to 10.6] | 2.30 [2.0 to 3.0] | 2.00 [2.0 to 2.0]

28. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum HAI Antibodies to PIV3 Day 28 Post Dose 1
Description: as for outcome 27
Time Frame: Day 28-34 after Dose 1 (Dose 1 was on Day 0)
Population: as for outcome 23
Measure: Mean (95% Confidence Interval); unit: GMT
Arm/Group | 10^4 MEDI-534 | 10^4 Placebo | 10^5 MEDI-534 | 10^5 Placebo | 10^6 MEDI-534 | 10^6 Placebo
Number analyzed (Participants) | 11 | 5 | 7 | 5 | 10 | 5
GMT | 13.24 [6.2 to 28.2] | 2.00 [2.0 to 2.0] | 19.50 [7.2 to 52.5] | 3.03 [2.0 to 7.0] | 14.93 [6.5 to 34.3] | 2.00 [2.0 to 2.0]

29. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum HAI Antibodies to PIV3 Day 28 Post Dose 2
Description: as for outcome 27
Time Frame: Day 28-34 after Dose 2 (Dose 2 was on Day 48-64)
Population: as for outcome 23
Measure: Mean (95% Confidence Interval); unit: GMT
Arm/Group | 10^4 MEDI-534 | 10^4 Placebo | 10^5 MEDI-534 | 10^5 Placebo | 10^6 MEDI-534 | 10^6 Placebo
Number analyzed (Participants) | 10 | 4 | 5 | 6 | 9 | 5
GMT | 13.93 [7.4 to 26.0] | 2.00 [2.0 to 2.0] | 24.25 [10.6 to 55.7] | 4.00 [2.0 to 8.0] | 11.76 [5.9 to 23.5] | 2.00 [2.0 to 2.0]

30. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum HAI Antibodies to PIV3 Day 28 Post Dose 3
Description: as for outcome 27
Time Frame: Day 28-34 after Dose 3 (Dose 3 was 48-64 days after Dose 2)
Population: as for outcome 23
Measure: Mean (95% Confidence Interval); unit: GMT
Arm/Group | 10^4 MEDI-534 | 10^4 Placebo | 10^5 MEDI-534 | 10^5 Placebo | 10^6 MEDI-534 | 10^6 Placebo
Number analyzed (Participants) | 10 | 3 | 5 | 5 | 8 | 4
GMT | 18.38 [10.6 to 32.0] | 2.00 [2.0 to 2.0] | 16.00 [7.0 to 36.8] | 3.03 [2.0 to 7.0] | 38.05 [17.4 to 107.6] | 2.00 [2.0 to 2.0]

31. Secondary Outcome: Number of Participants With Seroresponse to RSV 28 Days After Dose 1
Description: Seroresponse is equal to or greater than a 4-fold rise in RSV antibody from baseline as measured by microneutralization assay.
Time Frame: Days 28-34 after Dose 1 (Dose 1 was on Day 0)
Population: The immunogenicity population included all subjects who received investigational product and had valid results from serum samples obtained for immunogenicity evaluation for RSV.
Measure: Number; unit: participants
Arm/Group | 10^4 MEDI-534 | 10^4 Placebo | 10^5 MEDI-534 | 10^5 Placebo | 10^6 MEDI-534 | 10^6 Placebo
Number analyzed (Participants) | 11 | 5 | 7 | 4 | 9 | 5
participants | 2 | 0 | 3 | 0 | 4 | 0

32. Secondary Outcome: Number of Participants With Seroresponse to RSV 28 Days After Dose 2
Description: as for outcome 31
Time Frame: Days 28-34 after Dose 2 (Dose 2 was on Day 48-64)
Population: as for outcome 31
Measure: Number; unit: participants
Arm/Group | 10^4 MEDI-534 | 10^4 Placebo | 10^5 MEDI-534 | 10^5 Placebo | 10^6 MEDI-534 | 10^6 Placebo
Number analyzed (Participants) | 10 | 5 | 5 | 5 | 9 | 5
participants | 1 | 0 | 1 | 0 | 5 | 0

33. Secondary Outcome: Number of Participants With Seroresponse to RSV 28 Days After Dose 3
Description: as for outcome 31
Time Frame: Days 28-34 after Dose 3 (Dose 3 was 48-64 days after Dose 2)
Population: as for outcome 31
Measure: Number; unit: participants
Arm/Group | 10^4 MEDI-534 | 10^4 Placebo | 10^5 MEDI-534 | 10^5 Placebo | 10^6 MEDI-534 | 10^6 Placebo
Number analyzed (Participants) | 8 | 4 | 5 | 4 | 8 | 4
participants | 3 | 1 | 1 | 0 | 4 | 0

34. Secondary Outcome: Number of Participants With Seroresponse to PIV3 28 Days After Dose 1
Description: Seroresponse is equal to or greater than a 4-fold rise in PIV3 antibody from baseline as measured by HAI assay.
Time Frame: Days 28-34 after Dose 1 (Dose 1 was on Day 0)
Population: The immunogenicity population included all subjects who received investigational product and had valid results from serum samples obtained for immunogenicity evaluation for PIV3. Hemagglutination inhibition antibody results obtained on or after detection of wild-type HPIV3 in culture were not considered valid.
Measure: Number; unit: participants
Arm/Group | 10^4 MEDI-534 | 10^4 Placebo | 10^5 MEDI-534 | 10^5 Placebo | 10^6 MEDI-534 | 10^6 Placebo
Number analyzed (Participants) | 11 | 5 | 7 | 4 | 10 | 5
participants | 6 | 0 | 5 | 0 | 8 | 0

35. Secondary Outcome: Number of Participants With Seroresponse to PIV3 28 Days After Dose 2
Description: Seroresponse is equal to or greater than a 4-fold rise in PIV3 antibody from baseline as measured by HAI assay.
Time Frame: Days 28-34 after Dose 2 (Dose 2 was on Day 48-64)
Population: as for outcome 34
Measure: Number; unit: participants
Arm/Group | 10^4 MEDI-534 | 10^4 Placebo | 10^5 MEDI-534 | 10^5 Placebo | 10^6 MEDI-534 | 10^6 Placebo
Number analyzed (Participants) | 10 | 4 | 5 | 5 | 9 | 5
participants | 6 | 0 | 4 | 0 | 7 | 0

36. Secondary Outcome: Number of Participants With Seroresponse to PIV3 28 Days After Dose 3
Description: Seroresponse is equal to or greater than a 4-fold rise in PIV3 antibody from baseline as measured by HAI assay.
Time Frame: Days 28-34 after Dose 3 (Dose 3 was 48-64 days after Dose 2)
Population: as for outcome 34
Measure: Number; unit: participants
Arm/Group | 10^4 MEDI-534 | 10^4 Placebo | 10^5 MEDI-534 | 10^5 Placebo | 10^6 MEDI-534 | 10^6 Placebo
Number analyzed (Participants) | 10 | 3 | 5 | 4 | 8 | 4
participants | 8 | 0 | 3 | 0 | 8 | 0

ADVERSE EVENTS:
Time Frame: AEs:0-28 Days Postdose1, Postdose2, or postdose3 SAEs:0-180 Days Post Final Dose or Through 01 April Following Dosing for Sites in the USA, Whichever was Later
Arm/Group | 10^4 MEDI-534 | 10^4 PLACEBO | 10^5 MEDI-534 | 10^5 PLACEBO | 10^6 MEDI-534 | 10^6 PLACEBO
Serious Adverse Events (participants affected / at risk) | 1/13 | 0/6 | 0/9 | 1/6 | 0/10 | 0/5
Other Adverse Events (participants affected / at risk) | 11/13 | 5/6 | 8/9 | 5/6 | 9/10 | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10^4 MEDI-534 (N=13) | 10^4 PLACEBO (N=6) | 10^5 MEDI-534 (N=9) | 10^5 PLACEBO (N=6) | 10^6 MEDI-534 (N=10) | 10^6 PLACEBO (N=5)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10^4 MEDI-534 (N=13) | 10^4 PLACEBO (N=6) | 10^5 MEDI-534 (N=9) | 10^5 PLACEBO (N=6) | 10^6 MEDI-534 (N=10) | 10^6 PLACEBO (N=5)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Middle ear effusion (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tympanic membrane disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Tympanic membrane hyperaemia (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (2)
Eye discharge (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Eye disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eyelid margin crusting (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (8) | 3 (4) | 3 (6) | 2 (2) | 2 (2) | 1 (1)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infantile spitting up (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Teething (Gastrointestinal disorders) | 6 (13) | 0 (0) | 3 (5) | 2 (2) | 2 (4) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 2 (2) | 3 (5) | 4 (6) | 0 (0) | 1 (2)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body tinea (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Croup infectious (Infections and infestations) | 1 (2) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 1 (2) | 2 (2) | 1 (2)
Otitis media acute (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Roseola (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin candida (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Viral rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 1 (2) | 1 (1) | 3 (4) | 1 (1) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased activity (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Middle insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (5) | 2 (4) | 1 (2) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it is understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.